CLINICAL TRIAL: NCT00504179
Title: The Effect of Osteopathic Manipulative Treatment on Post-Operative Medical and Functional Recovery of Coronary Artery Bypass Graft Patients
Brief Title: The Effect of Osteopathic Manipulative Treatment on Recovery of Coronary Bypass Patients
Acronym: CABGOMT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Michigan State University (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: WIETING061855
Record Dates: First submitted 2007-07-17; First posted 2007-07-19 (Estimated); Last update posted 2007-07-19 (Estimated); Status verified 2007-07

CONDITIONS: Cardiovascular Disease
Keywords: coronary artery bypass graft; osteopathic manipulative treatment; cardiovascular disease
MeSH Terms: conditions — Cardiovascular Diseases | interventions — Manipulation, Osteopathic

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Procedure: Osteopathic Manipulative Treatment

SUMMARY:
The purpose of the study was to determine the effect on recovery after surgery of patients who received a standardized daily protocol of osteopathic manipulative treatment.Patients undergoing elective coronary artery bypass surgery were voluntarily enrolled in the study and assigned to one of three groups.One group received a standardized daily treatment protocol along with conventional care, another received daily similar placebo treatment with conventional care, and a final group received only conventional post surgical care.The research hypothesis was that daily treatment with osteopathic manipulative treatment would reduce hospital stay and hasten recovery from surgery.Persons in the treatment group had earlier discharge, and faster recovery of bowel function and basic mobility.

DETAILED DESCRIPTION:
Fifty-three persons were voluntarily enrolled into this randomized, double-blinded placebo controlled trial to examine the effects of osteopathic manipulative treatment (OMT) on the post operative recovery of persons undergoing elective coronary artery bypass graft (CABG) surgery. Participants were assigned randomly to one of three cohorts: one with only conventiobnal treatment, one with a daily standardized protocol of OMT and a third with a daily time matched placebo OMT protocol.All patients received standard state of the art care consistent with national standards of post CABG care. The study showed favorable trends in terms of hospital length of stay , return of bowel function, and mobility.

ELIGIBILITY:
Inclusion Criteria:

* Adults undergoing elective coronary artery bypass graft surgery who were patients of the same surgeon

Exclusion Criteria:

* prior coronary artery bypass graft procedure
* unstable psychiatric illness
* chronic pain
* open chest phenomenon
* unforeseen peri or postoperative complications

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 53 (Actual)
Dates: Start 2001-04; Study Completion 2005-10 (Actual)

PRIMARY OUTCOMES:
Recovery of mobility, bowel function, and reduced length of hospital stay.

CONTACTS AND LOCATIONS:
Overall Officials: Michael Wieting, Principal Investigator — Michigan State University
Locations (1):
- Ingham Regional Medical Center, Lansing, Michigan, United States